CLINICAL TRIAL: NCT01942785
Title: Interventional, Open-label, Flexible-dose, Exploratory Study of Brexpiprazole as Adjunctive Treatment of Irritability in Patients With Major Depressive Disorder and an Inadequate Response to Antidepressant Therapy
Brief Title: Study of Brexpiprazole as Adjunctive Treatment of Irritability in Patients With Major Depressive Disorder and an Inadequate Response to Antidepressant Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15353A
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder; Irritability
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental): Brexpiprazole adjunct to open-label commercially available Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI) antidepressant treatment (ADT)
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — 2-3 mg/day, once daily dose, tablets, for oral use. The patients received 1mg/day brexpiprazole during Week 1 and 2mg/day during Week 2 (up-titration) and from Weeks 3 to 6 they received 3mg/day; depending on tolerability the dose could be reduced to 2mg/day based on the investigator's judgement.

SUMMARY:
To explore the anti-impulsive and anti-aggressive properties of brexpiprazole in a naturalistic setting of depressed patients with irritability.

ELIGIBILITY:
Inclusion Criteria:

Main selection criteria at screening visit:

* The patient has a Major Depressive Episode (MDE) associated to Major Depressive Disorder (MDD) diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR™). The current MDE should be confirmed using the Mini International Neuropsychiatric Interview (MINI)
* The patient has an inadequate response to at least one antidepressant treatment (including the treatment the patient is taking at screening) in the current MDE, as documented by self-report as less than a pre-defined percentage response on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ).
* Pre-defined MADRS total score
* Pre-defined CGI-S total score
* The patient has had the current MDE for ≥10 weeks
* The patient is receiving a SSRI or SNRI antidepressant treatment for ≥6 weeks, at same dosage for ≥2 weeks
* Pre-defined Inventory of Depressive Symptomatology - Clinician-Rated - 30 items (IDS-C 30) Item 6 Mood (irritable) score

Main inclusion criteria at baseline visit:

* The patient still fulfils DSM-IV-TR™ criteria for MDE
* Pre-defined MADRS total score
* Pre-defined CGI-I (Lead-in period) score
* The patient received the same SSRI or SNRI antidepressant treatment at adequate doses during the entire lead-in period
* The patient has less than a pre-defined percentage decrease in MADRS score at the end of the lead-in period as compared to the screening visit
* The patient still has the pre-defined IDS-C 30 Item 6 Mood (Irritable) score

Exclusion Criteria:

* The patient has any current psychiatric disorder or Axis I disorder (DSM-IV-TR™ criteria), established as the principal diagnosis, other than MDD. All anxiety disorders, impulse-control disorders such as intermittent explosive disorder, as well as non-suicidal self-injury are not excluded diagnoses as far as they are not considered as principal diagnosis.
* The patient has a current Axis II (DSM-IV-TR™) diagnosis of antisocial, borderline, paranoid, schizoid, schizotypical, or histrionic personality disorder.
* The patient has experienced/experiences hallucinations, delusions, or any psychotic symptomatology in the current MDE.
* The patient, in the opinion of the investigator or based on C-SSRS rating, is at significant risk of suicide.
* The patient has started formal cognitive or behavioural therapy or systematic psychotherapy within 6 weeks prior to screening, or plans to start such therapy during the study. Any ongoing formal psychotherapy initiated more than 6 weeks prior to screening should be continued with the same methodology and at the same frequency and intensity during the entire study.
* The patient has a current diagnosis or history of substance abuse or dependence (excluding nicotine or caffeine) or alcohol abuse or dependence (DSM-IV-TR™ criteria) <6 months prior to the Screening Visit.
* The patient reports adjunctive treatment with an antipsychotic medication together with an antidepressant for 3 weeks or more during the current MDE.
* The patient has received electroconvulsive therapy (ECT) <6 months prior to the Screening Visit or at any time during the current MDE (if its duration is longer than 6 months).
* The patient has had vagus nerve stimulation or a deep brain stimulation device implanted for the management of depression.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (15):
- United States (15):
  - US015, Tucson, Arizona
  - US019, Glendale, California
  - US016, Oakland, California
  - US014, San Diego, California
  - US011, Denver, Colorado
  - US018, Hallandale, Florida
  - US009, Jacksonville, Florida
  - US005, Orlando, Florida
  - US006, Gaithersburg, Maryland
  - US012, Weymouth, Massachusetts
  - US003, Jamaica, New York
  - US001, Dayton, Ohio
  - US007, Portland, Oregon
  - US004, Memphis, Tennessee
  - US002, Seattle, Washington

REFERENCES:
- [Derived] Fava M, Menard F, Davidsen CK, Baker RA. Adjunctive Brexpiprazole in Patients With Major Depressive Disorder and Irritability: An Exploratory Study. J Clin Psychiatry. 2016 Dec;77(12):1695-1701. doi: 10.4088/JCP.15m10470. PMID 27379823

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 55 patients enrolled, only 54 were exposed to IMP and therefore included in the all-patients-treated set (APTS)
Groups:
- Brexpiprazole: Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant treatment (ADT) Brexpiprazole: 2-3 mg/day, once daily, tablets, for oral use
Period: Overall Study
Arm/Group | Brexpiprazole
Started | 54
Completed | 50
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The all-patients-treated set (APTS) comprises all patients who took at least one dose of brexpiprazole.
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.41 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 17
  White | 33
  More than one race | 0
  Unknown or Not Reported | 2
MADRS total score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS), n=54
  units on a scale | 28.52 (4.51)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). The overall number of baseline participants was based on the FAS, n=54
  units on a scale | 4.09 (0.40)
IDS-C30 item 6 score [Mean (Standard Deviation); unit: units on a scale] — The 30-item Inventory of Depressive Symptomatology - Clinician-Rated (IDS-C30) is a clinician-rated scale designed to assess the severity of depressive symptoms. The IDS-C30 item 6 measures mood (irritable) and is rated on a 4-point anchored scale from 0 (least severe) to 3 (most severe) with higher values indicating worse outcome. The overall number of baseline participants was based on the FAS, n=54
  units on a scale | 2.20 (0.41)
BIS-11 total score [Mean (Standard Deviation); unit: units on a scale] — The Barratt Impulsiveness Scale, Version 11 (BIS-11) is a patient-rated scale designed to assess impulsive personality traits. The BIS-11 consists of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). The total score ranges from 30 to 120 with higher values indicating worse outcome. The overall number of baseline participants was based on the FAS, n=54
  units on a scale | 73.20 (12.82)
KSQ anger-hostility score [Mean (Standard Deviation); unit: units on a scale] — The Kellner Symptom Questionnaire (KSQ) is a patient-rated scale designed to assess distress using symptoms of depression, anxiety, anger-hostility, and somatization. The KSQ anger-hostility subscale score ranges from 0 to 23 with higher values indicating worse outcome. The overall number of baseline participants was based on the FAS, n=54
  units on a scale | 14.83 (4.78)
AAQ anger attacks [Number; unit: participants] — The Anger Attacks Questionnaire (AAQ) is a patient-rated scale designed to assess the presence of anger attacks. The AAQ consists of 7 items. Patients are classified as having anger attacks when exhibiting the following 4 criteria: 1) irritability, 2) overreaction to minor annoyances, 3) occurrence of anger attacks (at least one of which occurred within the period), and 4) experienced 4 or more specific symptoms during at least one of the attacks. The overall number of baseline participants was based on the FAS, n=54
  participants
    no | 37
    yes | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in SIS Total Score
Description: The Sheehan Irritability Scale (SIS) is a patient-rated scale designed to measure irritability. The SIS consists of 7 subscales assessing irritability, frustration, edginess/impatience/overreaction, moodiness, anger with self, anger with others, and temper. The subscales are summarised to give the total score which ranges from 0 to 70, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -21.13 (2.55)

2. Primary Outcome: Change From Baseline to Week 6 in SIS Item 1 Score
Description: The Sheehan Irritability Scale (SIS) is a patient-rated scale designed to measure irritability. The SIS item 1 assess how much the patient has suffered from irritability in the past week. The SIS item 1 ranged from 0 to 10 with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -3.45 (0.36)

3. Primary Outcome: Change From Baseline to Week 6 in IDS-C30 Item 6 Score
Description: The 30-item Inventory of Depressive Symptomatology - Clinician-Rated (IDS-C30) is a clinician-rated scale designed to assess the severity of depressive symptoms. The IDS-C30 item 6 measures mood (irritable) and is rated on a 4-point anchored scale from 0 (least severe) to 3 (most severe) with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -1.22 (0.13)

4. Primary Outcome: Change From Baseline to Week 6 in Delay Discounting - Log-transformed MCQ Scores
Description: The Monetary Choice Questionnaire (MCQ) is a patient-completed questionnaire designed to measure delay discounting, an index of impulsive behaviour. The MCQ consists of 27 choices between immediate and delayed rewards. The patients choose repeatedly between two hypothetical sums of money: a smaller amount now or a larger amount in the future (for example, ''Would you prefer $27 today or $50 in 21 days?"). The answers provide an estimate of the patient's discounting rate. The discounting rate parameter takes values between 0 and 1 and higher discounting rates indicate impulsivity. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: log-transformed units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
log-transformed units on a scale | 0.00 (0.24)

5. Primary Outcome: Change From Baseline to Week 6 in BIS-11 Total Score
Description: The Barratt Impulsiveness Scale, Version 11 (BIS-11) is a patient-rated scale designed to assess impulsive personality traits. The BIS-11 consists of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). The total score ranges from 30 to 120 with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -4.85 (0.86)

6. Primary Outcome: Change From Baseline to Week 6 in KSQ Anger-hostility Subscore
Description: The Kellner Symptom Questionnaire (KSQ) is a patient-rated scale designed to assess distress using symptoms of depression, anxiety, anger-hostility, and somatization. The KSQ anger-hostility subscale score ranges from 0 to 23 with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -7.72 (0.92)

7. Primary Outcome: Shift From Baseline to Week 6 in Anger Attacks (AAQ)
Description: The Anger Attacks Questionnaire (AAQ) is a patient-rated scale designed to assess the presence of anger attacks over a period of time. The AAQ consists of 7 items. Patients are classified as having anger attacks when exhibiting the following 4 criteria: 1) irritability, 2) overreaction to minor annoyances, 3) occurrence of anger attacks (at least one of which occurred within the period), and 4) experienced 4 or more specific symptoms during at least one of the attacks. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS) and OC. Only patients who have both baseline and Week 6 data observed were included; the number of participants analysed is therefore smaller than the defined FAS.
Measure: Number; unit: participants
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 50
participants
  no to no | 28
  no to yes | 5
  yes to no | 15
  yes to yes | 2

8. Primary Outcome: Change From Baseline to Week 6 in IDS-C30 Total Score
Description: The 30-item Inventory of Depressive Symptomatology - Clinician-Rated (IDS-C30) is a clinician-rated scale designed to assess the severity of depressive symptoms. The IDS-C30 consists of 30 items assessing the symptoms of depression, as well as commonly associated symptoms (for example, anxiety, irritability), and topics relevant to melancholic or atypical features; the patient rates only one of the 2 items assessing appetite (decreased or increased), and only one of the 2 items assessing weight (loss or gain). Each of the items is rated on a 4-point anchored scale from 0 (least severe) to 3 (most severe). The total score is the sum of the 28 scored items, and ranges from 0 to 84, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -17.81 (1.57)

9. Primary Outcome: Change From Baseline to Week 6 in KSQ Depression Subscore
Description: The Kellner Symptom Questionnaire (KSQ) is a patient-rated scale designed to assess distress using symptoms of depression, anxiety, anger-hostility, and somatization. The KSQ depression subscale score ranges from 0 to 23, with higher values indicating worse outcome . As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -7.70 (0.93)

10. Primary Outcome: Change From Baseline to Week 6 in MADRS Total Score
Description: The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -14.19 (1.27)

11. Primary Outcome: Change From Baseline to Week 6 in CPFQ Total Score
Description: The Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) is a patient-rated scale designed to assess cognitive and executive dysfunction including symptoms of fatigue in mood and anxiety disorders. The CPFQ consists of 7 items, each rated on a scale from 1 (greater than normal functioning) to 6 (poorer than normal functioning). The total score of the 7 items ranges from 7 to 42, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -7.72 (0.97)

12. Primary Outcome: Change From Baseline to Week 6 in CGI-S Score
Description: The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -1.43 (0.16)

13. Primary Outcome: CGI-I Score at Week 6
Description: The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 6
Population: Full-analysis set (FAS), this endpoint presents descriptive statistics for CGI-I based on patients who have CGI-I score observed at Week 6; the number of participants analysed is therefore smaller than the defined FAS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 50
units on a scale | 2.18 (0.16)

14. Primary Outcome: Change From Baseline to Week 6 in KSQ Total Score
Description: The Kellner Symptom Questionnaire (KSQ) is a patient-rated scale designed to assess distress using symptoms of depression, anxiety, anger-hostility, and somatization. The KSQ consists of 92 items which form the basis for the four subscales: depression, anxiety, anger-hostility, and somatic; of which 68 items indicate symptoms (symptom subscales) and 24 items are antonyms of some of the symptoms and indicate well-being (well-being subscales). A "yes" or "true" response on the symptom subscales scores 1, and a "no" or "false" on the well-being subscales scores 1. The maximum score for each symptom subscale is 17, and the maximum score for each well-being subscale is 6. The score of each subscale ranges from 0 to 23 (the sum of the symptom subscale and the well-being subscale). A higher score indicates more distress. The total score ranges from 0 to 92. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale | -24.36 (2.94)

15. Primary Outcome: Change From Baseline to Week 6 in Delay Discounting - Log-transformed EDT DPDT Scores
Description: DPDT consists of approximately 110 choices between an immediate reward or a higher delayed reward, and between an immediate reward or a higher reward that only comes with a certain probability. The tasks are scored independently of each other and do not yield a total score. There will be two derived variables from this task; a delayed discounting rate and a probability discounting rate. The delay discounting value takes values from 0 and up, a higher delay discounting value indicates greater impulsivity. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: full-analysis set (FAS). Only patients who have observed data at Week 6 were included in the ANCOVA analysis; the number of participants analysed is therefore smaller than the defined FAS.
Measure: Mean (Standard Error); unit: log transformed units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
log transformed units on a scale
  DPDT delay score | -0.223 (0.349)
  DPDT Probability Score | -0.295 (0.271)

16. Primary Outcome: Change From Baseline to Week 6 in Delay Discounting - EDT DRT Score
Description: DRT consists of 60 choices between an immediate reward or a higher delayed reward. The number of impulsive choices will be a continuous variable estimated from how many immediate choices based on 60 possible. The number ranges between 0 and 60, with a higher value indicating more impulsivity. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: as for outcome 15
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
units on a scale | 0.74 (1.97)

17. Primary Outcome: Change From Week 6 to Week 10 in SIS Total Score
Description: The Sheehan Irritability Scale (SIS) is a patient-rated scale designed to measure irritability. The SIS consists of 7 subscales assessing irritability, frustration, edginess/impatience/overreaction, moodiness, anger with self, anger with others, and temper. The patient rates the extent to which they have suffered from these symptoms. Each subscale has verbal descriptors (not at all, mildly, moderately, markedly, and extremely) as well as numerical scores from 0 (not at all) to 10 (extremely) that provide more precise levels of the verbal descriptors. One additional question assesses number of days impaired by irritability over the period. The subscales are summarised to give the total score which ranges from 0 to 70, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 6 and Week 10
Population: Completer's-analysis set (CAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 48
units on a scale | 4.4 (2.4)

18. Primary Outcome: Change From Week 6 to Week 10 in SIS Item 1 Score
Description: The Sheehan Irritability Scale (SIS) is a patient-rated scale designed to measure irritability. The SIS item 1 assess how much the patient has suffered from irritability in the past week, using verbal descriptors (not at all, mildly, moderately, markedly, and extremely) as well as numerical scores from 0 (not at all) to 10 (extremely) that provide more precise levels of the verbal descriptors. The SIS item 1 ranged from 0 to 10 with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 6 and Week 10
Population: Completer's-analysis set (CAS). Only patients who have observed data at Week 10 were included in the ANCOVA analysis; the number of participants analysed is therefore smaller than the defined CAS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
units on a scale | 0.5 (0.4)

19. Primary Outcome: Change From Week 6 to Week 10 in Delay Discounting - MCQ Scores
Description: as for outcome 4
Time Frame: Week 6 and Week 10
Population: as for outcome 18
Measure: Mean (Standard Error); unit: log-transformed units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
log-transformed units on a scale | 0.35 (0.15)

20. Primary Outcome: Change From Week 6 to Week 10 in BIS-11 Total Score
Description: The Barratt Impulsiveness Scale, Version 11 (BIS-11) is a patient-rated scale designed to assess impulsive personality traits. The BIS-11 consists of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). The scores provide information to assess 6 first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and 3 second-order factors (motor impulsiveness, non-planning impulsiveness, and attentional impulsiveness). The total score ranges from 30 to 120 with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 6 and Week 10
Population: Completer's-analysis set (CAS). Only patients who have observed data at Week 10 were included in the ANCOVA analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 47
units on a scale | -1.2 (0.9)

21. Primary Outcome: Change From Week 6 to Week 10 in KSQ Anger-hostility Subscore
Description: as for outcome 6
Time Frame: Week 6 and Week 10
Population: Completer's-analysis set (CAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 48
units on a scale | 1.2 (1.0)

22. Primary Outcome: Change From Week 6 to Week 10 in KSQ Depression Subscore
Description: as for outcome 9
Time Frame: Week 6 and Week 10
Population: Completer's-analysis set (CAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 48
units on a scale | 2.1 (1.0)

23. Primary Outcome: Change From Week 6 to Week 10 in CGI-S Score
Description: as for outcome 12
Time Frame: Week 6 and Week 10
Population: Completer's-analysis set (CAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 48
units on a scale | 0.3 (0.1)

24. Primary Outcome: Change From Baseline to Week 6 in MADRS Total Score in Patients With a Pre-defined Baseline BIS-11 Total Score
Description: The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. Subgroup analyses were performed for the change from Baseline to Week 6 in MADRS total score based on the patients' BIS-11 total score at Baseline. The subgroups denoted BIS-11_HIGH had a BIS-11 total score at Baseline ≥median at baseline and the subgroups denoted BIS-11_LOW had a BIS-11 total score <median at baseline. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Brexpiprazole: Brexpiprazole adjunct to open-label commercially available Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI) antidepressant treatment (ADT)
  Brexpiprazole:2-3 mg/day, once daily dose, tablets, for oral use
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale
  BIS-11_HIGH (n=27) | -14.41 (1.71)
  BIS-11_LOW (n=27) | -15.45 (1.78)

25. Primary Outcome: Change From Baseline to Week 6 in CGI-S Score in Patients With a Pre-defined Baseline BIS-11 Total Score
Description: The subgroups denoted BIS-11_HIGH had a BIS-11 total score at Baseline ≥median at baseline and the subgroups denoted BIS-11_LOW had a BIS-11 total score <median at baseline. The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 6
Population: full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Brexpiprazole: Brexpiprazole adjunct to open-label commercially available Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI) antidepressant treatment (ADT)
  Brexpiprazole: 2-3 mg/day, once daily dose, tablets, for oral use
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale
  BIS-11_HIGH (n=27) | -1.31 (0.21)
  BIS-11_LOW (n=27) | -1.53 (0.20)

26. Primary Outcome: CGI-I Score at Week 6 Patients With a Pre-defined Baseline BIS-11 Total Score
Description: The subgroups denoted BIS-11_HIGH had a BIS-11 total score at Baseline ≥median at baseline and the subgroups denoted BIS-11_LOW had a BIS-11 total score <median at baseline. The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 6
Population: full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 54
units on a scale
  BIS-11_HIGH (n=27) | 2.48 (0.23)
  BIS-11_LOW (n=23) | 1.83 (0.20)

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (week 6)
Description: Treatment-Emergent Adverse Events
Arm/Group | Brexpiprazole
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 31/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=54)
Diarrhoea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Fall (Injury, poisoning and procedural complications) | 3
Weight increased (Investigations) | 3
Increased appetite (Metabolism and nutrition disorders) | 4
Akathisia (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No